CLINICAL TRIAL: NCT01530373
Title: A Phase II Randomized Study of Solifenacin Compared to Clonidine for Reducing Hot Flashes Among Breast Cancer Patients Receiving Adjuvant Hormonal Therapy
Brief Title: Solifenacin Compared to Clonidine for Reducing Hot Flashes Among Breast Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 132500
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hot Flashes; Breast Cancer
Keywords: hot flashes; breast cancer; aromatase inhibitors; solifenacin; clonidine; quality of life
MeSH Terms: conditions — Hot Flashes; Breast Neoplasms | interventions — Solifenacin Succinate; Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- solifenacin (Experimental): oral solifenacin 5.0 mg daily for 3 weeks
  Interventions: Drug: solifenacin
- clonidine (Active Comparator): oral clonidine 0.1 mg daily for 3 weeks
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: solifenacin — oral solifenacin 5.0 mg daily for 3 weeks
  Other Names: Vesicare
  Arms: solifenacin
Drug: Clonidine — oral clonidine 0.1 mg daily for 3 weeks
  Other Names: Catapres, Dixarit
  Arms: clonidine

SUMMARY:
Hot flashes present a considerable problem for many breast cancer patients; these symptoms may be intensified by hormonal therapies, such as aromatase inhibitors or tamoxifen. This study examines the value of solifenacin (a muscarinic acetylcholine receptor antagonist) in reducing hot flashes, compared with clonidine (a medication often used for treating hot flashes).

DETAILED DESCRIPTION:
There has been considerable interest in developing new treatment strategies for managing hot flashes among women with breast cancer, in view of the limitations associated with currently available treatments. This randomized study evaluates the safety and efficacy of 3 weeks of solifenacin compared to 3 weeks of clonidine, for women receiving adjuvant hormonal therapy (aromatase inhibitors or tamoxifen) for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of invasive breast cancer or DCIS
* Currently taking aromatase inhibitors or tamoxifen
* Not receiving hormone replacement therapy for minimum of one month
* Age 18 years or older
* Self-reported hot flashes at least fourteen times per week
* Self-reported hot flashes for at least one month
* If receiving non-tricyclic antidepressants (venlafaxine, paroxetine, citalopram, sertraline, etc.) or gabapentin, no change in regimen in past 4 weeks.

Exclusion Criteria:

* Receiving any other treatment for hot flashes within the past month, including estrogens, progestins, androgens, or gabapentin.
* Current use of clonidine or solifenacin. (If patients have been off of these for one month, then they are eligible)
* History of severe renal or moderate or severe hepatic impairment, as indicated by physical exam and medical record
* Concurrent or planned chemotherapy or radiotherapy (within next 3 months)
* Currently receiving tricyclic antidepressants, monoamine oxidase inhibitors, barbiturates, pimozide.
* Currently using CYP3A4 inducers (i.e., aminoglutethimide, carbamazepine, dexamethasone, efavirenz, ethosuximide, griseofulvin, modafinil, nafcillin, nevirapine, oxcarbazepine, phenobarbital, phenylbutazone, phenytoin, primidone, rifabutin, rifampin, rifapentine, St. John's Wort, sulfadimidine, sulfinpyrazone, troglitazone) or potent CYP3A4 inhibitors (i.e., chloramphenicol, clarithromycin, erythromycin, imatinib mesylate, indinavir sulfate, itraconazole, ketoconazole, nefazoldone, nelfinavir mesylate, ritonavir, telithromycin, troleandomycin).
* Uncontrolled or poorly controlled narrow-angle glaucoma, urinary retention, gastric retention (evaluated from history & physical exam and medical record)
* Hypotension or uncontrolled hypertension (160/95 > BP < 100/60)
* Severe coronary insufficiency, conduction disturbances, recent myocardial infarction (within past 3 months), cerebrovascular disease, syncope (evaluated from history & physical and medical record)
* History of allergy or adverse reactions to clonidine or solifenacin
* ECOG status > 2 (in bed more than 50% of day)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2012-02; Primary Completion 2026-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy: hot flash composite and frequency scores (daily diary) | from baseline to end of treatment (3 weeks)
  to evaluate changes in hot flash composite and frequency scores for women receiving 3 weeks of oral solifenacin compared to those receiving 3 weeks of oral clonidine
Safety: number of clinician-rated adverse events | from consent until end of study (approximately 9 weeks)
  to evaluate changes in number of adverse events for women receiving 3 weeks of oral solifenacin compared to those receiving 3 weeks of oral clonidine

SECONDARY OUTCOMES:
daily functioning (Hot Flash-Related Daily Interference score) | from baseline to end of treatment (3 weeks)
  to evaluate changes in daily functioning (Hot Flash-Related Daily Interference Score) for women receiving 3 weeks of oral solifenacin compared to those receiving 3 weeks of oral clonidine
sleep (Insomnia Severity Index) | from baseline to end of treatment (3 weeks)
  To evaluate changes in sleep
quality of life (Illness Cognition Questionnaire, SF-12) | from baseline to end of treatment (3 weeks)
  to evaluate changes in health-related quality of life. (Additional analyses will be observational, exploring associations between quality of life and meaning-making.)

CONTACTS AND LOCATIONS:
Overall Officials: Allen C Sherman, PhD, Principal Investigator — Universitiy of Arkansas for Medical Sciences
Locations (1):
- Winthrop P. Rockefeller Cancer Institute, University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States